CLINICAL TRIAL: NCT05040724
Title: Evaluation of the Impact of the Administration of Single Dose of Ivermectin in the Early Phase of COVID-19 on the Time to Negativation of the SARS-COV-2 Viral Load Determinated by RT-PCR
Brief Title: Evaluation of the Impact of the Administration of Single Dose of Ivermectin in the Early Phase of COVID-19
Acronym: IVERCoV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Raincy Montfermeil Hospital Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-005423-37
Record Dates: First submitted 2021-09-09; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-06

CONDITIONS: To Assess the Reduction in the Viral Load of SARS-CoV-2 in Patients Receiving Ivermectin Compared to Those Receiving Standard Care
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, double-blind, randomized trial in two parallel groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized into one of two groups in a 1: 1 ratio The randomization will be centralized and carried out electronically by IWRS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (Experimental): Ivermectin 3mg, on tablet. As a single dose of 400 µg / kg orally (rounded down to the nearest unit). T+ usual care
  Interventions: Drug: Ivermectin
- control (Placebo Comparator): placebo of ivermectin administered in the same manner as the active drug in experimental arm + usual care
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — ivermectin placebo
  Other Names: placebo

SUMMARY:
The action of ivermectin in vitro on the viral replication of SARS-CoV-2 was demonstrated and published by an Australian team in June 2020. On the other hand, the doses to be administered in vivo to reach the concentrations described in vitro would lead to toxicities especially neurological, in treated patients, . However, some trials and studies, such as the ICON3 study, demonstrate the clinical efficacy of ivermectin administered at lower doses (200 µg / kg) in hospitalized patients with COVID-19.

The use of ivermectin in the early stages of the disease has not yet been studied. The administration of the maximum authorized dose (MA) of ivermectin could at least slow down the replication of the virus in vivo before the inflammatory phase of COVID-19, and reduce the duration of symptoms as well as the risk of hospitalization of patients, especially in critical care.

Unlike other studies conducted so far on COVID-19, IVERCoV will target the "viral" phase of the disease by screening patients in the city. In addition, home visits (symptom recording +/- PCR) will make it easier to monitor patients during the study.

DETAILED DESCRIPTION:
The action of ivermectin in vitro on viral replication of SARS-CoV-2 was demonstrated and published by an Australian team in June 2020. On the other hand, the doses to be administered in vivo making it possible to reach the concentrations described in vitro would result in toxicities in treated patients, especially neurological. However, some trials and studies, such as the ICON3 study, demonstrate the clinical efficacy of ivermectin administered at lower doses (200 µg / kg) in hospitalized patients with COVID-19.

The use of ivermectin in the early stages of the disease has not yet been studied. The administration of the maximum authorized dose (MA) of ivermectin could at least slow down the replication of the virus in vivo before the inflammatory phase of COVID-19, and reduce the duration of symptoms as well as the risk of hospitalization of patients, especially in critical care.

Unlike other studies conducted so far on COVID-19, IVERCoV will target the "viral" phase of the disease by screening patients in the city. In addition, home visits (symptom recording +/- PCR) will make it easier to monitor patients during the study.

Prospective, multicenter, double-blind, randomized trial in two parallel groups:

* a control group: with administration of a placebo in addition to the usual treatment
* an experimental group: treated with ivermectin 400 µg / kg in addition to the usual treatment.

The primary endpoint: negation of the RT-PCR test on nasopharyngeal samples of SARS-CoV-2 on D3 of taking Ivermectin compared to the control group (placebo).

The secondary endpoints are:

* Evolution of symptoms from D0 to D28,
* SARS-CoV-2 viral load negativation kinetics measured on D0, D3, D7, D14 after treatment by ivermectin,
* comparison of the number of RT-PCR amplification cycles (Ct: Cycle threshold) in each group,
* number of patients having recourse to home oxygen therapy,
* number of patients hospitalized and / or requiring oxygen therapy,
* number of patients admitted to intensive care,
* number of deaths.

  200 patients will be enrolled: 100 patients for each randomization group.

ELIGIBILITY:
Inclusion Criteria:

* patient ≥ 18 years old,
* symptomatic COVID-19 for less than 96 hours (see list of symptoms in appendix),
* tested positive for SARS-CoV-2 by RT-PCR on a nasopharyngeal sample within 48 hours of inclusion,
* following an effective method of contraception for women of childbearing age,
* affiliated to a social security scheme,
* informed and written consent from patient.

Exclusion Criteria:

* patient requiring normal hospitalization or intensive care
* oxygen-requiring patient,
* with a history of parasitosis, in particular filariasis,
* with a history of hypereosinophilia,
* notion of recent travel (less than 3 months) in poor hygienic conditions
* taking ivermectin in the last 12 months,
* contraindications to ivermectin or one of the constituents of the drug (known history of allergies),
* pregnant or breastfeeding women,
* participation in another interventional study relating to COVID-19 concerning a drug during this research,
* patient under AME or without social security coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
negativation of the RT-PCR test on nasopharyngeal samples of SARS-CoV-2 | Day 3
  negativation of the RT-PCR test on nasopharyngeal samples of SARS-CoV-2 on D3 of taking Ivermectin compared to the control group (placebo).

CONTACTS AND LOCATIONS:
Locations (1):
- GHI Le Raincy Montfermeil, Montfermeil, France